CLINICAL TRIAL: NCT00212394
Title: A Prospective, Epidemiological Study of the Incidence and Nature of Tourniquet Complications in Norway
Brief Title: Tourniquet Complications in Orthopaedic Surgery
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: ADOD1
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Tourniquet Complications; Paresis; Palsy; Nerve Compression
Keywords: Tourniquet; paresis
MeSH Terms: conditions — Paresis; Paralysis; Neuroma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of the study is to establish the number and nature of complications that we, the researchers, have with the use of a tourniquet in orthopaedic surgery in Norway.

DETAILED DESCRIPTION:
This is a multicenter, prospective study where contact persons in 10 different hospitals throughout Norway monitor problems and complications that occur in relation with tourniquet use in orthopaedic surgery. If a complication occurs, it is documented in detail by the contact person.

ELIGIBILITY:
Inclusion Criteria:

* All patients in 10 orthopaedic hospitals in Norway undergoing surgery which requires a tourniquet, from 1 january to 31 of december 2005

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2005-01 (Actual); Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vilhjalmur Finsen, Profesor, Study Director — National Taiwan Normal University
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Odinsson A, Finsen V. Tourniquet use and its complications in Norway. J Bone Joint Surg Br. 2006 Aug;88(8):1090-2. doi: 10.1302/0301-620X.88B8.17668. PMID 16877612